CLINICAL TRIAL: NCT04156646
Title: A Single-Center, Part-Randomized, Open-Label, Single-Dose, Three-Period, Crossover Study to Investigate the Effect of Esomeprazole and The Effect of Food on the Pharmacokinetics of Balovaptan in Healthy Volunteers
Brief Title: A Study to Investigate the Effect of Esomeprazole and the Effect of Food on the Pharmacokinetics of Balovaptan in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WP41047
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — balovaptan; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment sequence ABC (Experimental): In Period 1 participants will receive 1 tablet of balovaptan after high-fat, high-calorie meal. In Period 2, after 12 to 21 days wash-out, participants will receive 1 tablet of balovaptan after 10-hour fast. In Period 3 participants will receive esomeprazole administered once daily for 6 days and with a single oral dose of balovaptan in the fasted state 1 hour after the fifth esomeprazole dose
  Interventions: Drug: Balovaptan; Drug: Esomeprazole
- Treatment sequence BAC (Experimental): In Period 1 participants will receive 1 tablet of balovaptan after 10-hour fast. In Period 2, after 12 to 21 days wash-out, participants will receive 1 tablet of balovaptan after high-fat, high-calorie meal. In Period 3 participants will receive esomeprazole administered once daily for 6 days and with a single oral dose of balovaptan in the fasted state 1 hour after the fifth esomeprazole dose
  Interventions: Drug: Balovaptan; Drug: Esomeprazole

INTERVENTIONS:
Drug: Balovaptan — Balovaptan will be administered after a high-fat, high-calorie meal (Treatment A), after a 10-hour fast (Treatment B), and after a 10-hour fast with esomeprazole 40 mg (Treatment C)
Drug: Esomeprazole — Esomeprazole will be administered once daily for 6 days and with a single dose of balovaptan 1 hour after the fifth esomeprazole dose

SUMMARY:
This study will investigate the effect of food and the effect of esomeprazole on the pharmacokinetics (PK) of a single dose of balovaptan in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* No evidence of any active or chronic disease
* Body mass index (BMI) between 18 and 32 kg/m2 inclusive, at screening
* For women of childbearing potential: if engaging in heterosexual activity, agreement to use at least two adequate forms of contraception during the entire study and for 90 days following the last dose of study drug
* For men: agreement to use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* Pregnancy or lactation (positive serum pregnancy test at screening or at admission)
* Any condition or disease detected during the medical interview/physical examination that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the Investigator
* In the opinion of the Investigator, any major illness within 4 weeks prior to the screening examination or any febrile illness within 1 week prior to screening.
* History of any clinically significant, as determined by the investigator, gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological, lymphatic, musculoskeletal, genitourinary, immunological, dermatological, or connective tissue or allergic disease, metabolic disorder, or cancer
* Signs and symptoms potentially indicative of peripheral neuropathy
* History or evidence of any medical condition potentially altering the absorption, distribution, metabolism, or elimination of drugs
* A history of clinically significant in the opinion of the Investigator hypersensitivity
* History or presence of clinically significant ECG abnormalities before study drug administration
* Clinically significant abnormalities in laboratory test results
* History of coagulopathies, bleeding disorders, or blood dyscrasias
* Current suicidal risk, in the opinion of the Investigator
* Unexplained syncope during the 6 months prior to screening or with presyncopal and/or syncopal symptoms during orthostatic challenge testing
* Current smoker or user of tobacco or nicotine-containing products or subjects who have smoked or used tobacco or nicotine-containing products within 3 months prior to first study drug administration
* Suspicion of or presence of a clinically relevant history of or current alcohol and/or other substance abuse or addiction.
* Alcohol consumption of >14 units per week for males and females
* Positive urine alcohol test or urine drug screen at screening or Day -1 of any treatment period
* Hormone replacement therapy if postmenopausal status cannot be ascertained from medical history or FSH levels
* Clinically relevant deviation from normal in the physical examination including vital signs, as determined by the investigator
* Positive result for HIV 1, HIV 2, hepatitis C virus antibody, or hepatitis B core (HBc) antibody.
* Participation in an investigational drug or device study within 4 weeks or 5 times the elimination half-life, whichever is longer, prior to first dosing, or within 5 months prior to first administration of study drug in case of a study with a biological, as calculated from the day of Follow-up visit from the previous study
* Donation of blood or plasma or significant blood loss within 3 months prior to screening
* Dietary restrictions that would prohibit the consumption of standardized meals or the highfat, high-calorie meal planned for this study
* Use of any prohibited medications or food before study start or subjects who do not agree to refrain from consuming prohibited medications or food during the study
* Conditions requiring concomitant medication during the study (including for dental conditions).
* Any prescribed systemic or topical medication within 4 weeks (or within 5 times the elimination half-life of the medication, whichever is longer) of the first administration of study drug
* Used any nonprescribed systemic or topical medication or herbal remedies within 7 days before the first study drug administration
* Received any medications known to chronically alter drug absorption or elimination processes within 4 weeks before the first administration of study drug
* Use of any drugs or substances, including herbal treatments such as St John's wort, that are known to be substrates, inducers, or inhibitors of CYP3A4 within 4 weeks before the first administration of study drug
* Use of any drugs or substances, including herbal treatments, such as fluoxetine, fluvoxamine, aspirin, norethisterone, rifampicin, etc that are known to be substrates, inducers, or inhibitors of CYP2C19 within 4 weeks before the first administration of study drug
* Subjects under judicial supervision, guardianship, or curatorship
* Poor venous access for blood sampling
* Participants who are intolerant to sucrose
* Previous exposure to balovaptan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- PRA International Clinical Pharmacology Center (EDS US Clinic), Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening was conducted between Day -28 and Day -2.
Groups:
- Treatment Sequence ABC: Participants were randomized to ABC sequence on Day 1 of Period 1 with the treatments being as follows:
  * Treatment A: 20 mg balovaptan administered as a single oral dose following consumption of high-fat, high-calorie meal
  * Treatment B: 20 mg balovaptan administered as a single oral dose after a ≥10-hour fast
  * Treatment C: 40 mg esomeprazole administered once daily (QD) for 6 days and with a single dose of balovaptan 20 mg in the fasted state 1 hour after the fifth esomeprazole dose
- Treatment Sequence BAC: Participants were randomized to BAC sequence on Day 1 of Period 1 with the treatments being as follows:
  * Treatment B: 20 mg balovaptan administered as a single oral dose after a ≥10-hour fast
  * Treatment A: 20 mg balovaptan administered as a single oral dose following consumption of high-fat, high-calorie meal
  * Treatment C: 40 mg esomeprazole administered once daily (QD) for 6 days and with a single dose of balovaptan 20 mg in the fasted state 1 hour after the fifth esomeprazole dose
Period: Treatment Period 1 (6 Days)
Arm/Group | Treatment Sequence ABC | Treatment Sequence BAC
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Wash-out Period (12- to 21-days)
Arm/Group | Treatment Sequence ABC | Treatment Sequence BAC
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Treatment Period 2 (6 Days)
Arm/Group | Treatment Sequence ABC | Treatment Sequence BAC
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Wash-out Period (12- to 21-days)
Arm/Group | Treatment Sequence ABC | Treatment Sequence BAC
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Treatment Period 3 (6 Days)
Arm/Group | Treatment Sequence ABC | Treatment Sequence BAC
Started | 8 | 8
Completed | 8 | 7
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABC | Treatment Sequence BAC | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (11.96) | 47.1 (13.26) | 43.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Balovaptan
Description: Maximum plasma concentration of Balovaptan is estimated using non-compartmental methods. Observed peak analyte concentration obtained directly from the experimental data without interpolation, expressed in concentration units
Time Frame: Samples at predose, and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 144, and 192 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Balovaptan 20 mg Fed: Single oral doses of balovaptan 20 mg (1 × 20 mg tablet) were administered following consumption of a high-fat, high-calorie meal (Treatment A).
- Balovaptan 20 mg Fasted: Single oral doses of balovaptan 20 mg (1 × 20 mg tablet) were after a ≥ 10 h fast (Treatment B)
- Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted: Single oral doses of balovaptan 20 mg (1 × 20 mg tablet) were coadministered with esomeprazole 40 mg (Treatment C) in a fasted state
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
ng/mL | 74.83 (42.6) | 97.44 (44.6) | 79.67 (38.3)

2. Primary Outcome: Mean Area Under the Concentration-Time Curve From Time Extrapolated to Infinity (AUC (0-inf)) of Balovaptan
Description: Area under the plasma concentration-time curve (time 0 to infinity) of Balovaptan is estimated using non-compartmental methods from the concentration-time profiles. Percent extrapolation less than or equal to 20% is required to obtain a reliable AUC0-inf.
Time Frame: as for outcome 1
Population: For one participant with Balovaptan 20 mg Fasted+ Esomeprazole 40 mg Fasted, AUC(0-inf)%extrap was > 20%, so AUC(0-inf) and T1/2 were not included in summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 15
h*ng/mL | 1736.7 (51.3) | 1705.7 (55.9) | 1820.0 (46.9)

3. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to 24 Hours (AUC(0-24h)) of Balovaptan
Description: Area under the plasma concentration-time curve of Balovaptan from time 0 to 24 hours post-dose is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: Samples at predose, and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16 and 24 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h*ng/mL | 935.2 (31.7) | 945.2 (30.8) | 965.0 (30.7)

4. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Balovaptan
Description: Area under the concentration-time curve (time 0 to time of last quantifiable concentration) of Balovaptan is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h*ng/mL | 1671.0 (50.2) | 1636.1 (53.3) | 1650.9 (48.3)

5. Primary Outcome: Time to Reach Cmax in Plasma (Tmax) of Balovaptan
Description: Time to maximum plasma concentration of Balovaptan is defined as first observed time to reach peak analyte concentration obtained directly from the experimental data without interpolation, expressed in time units and estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h | 4.50 [0.50 to 8.00] | 1.00 [0.50 to 3.00] | 1.75 [1.00 to 4.00]

6. Primary Outcome: Last Quantifiable Concentration (Clast) of Balovaptan
Description: Last quantifiable concentration is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
ng/mL | 1.693 (45.2) | 1.745 (57.3) | 2.253 (142.8)

7. Primary Outcome: Time To the Last Quantifiable Concentration (Tlast) of Balovaptan
Description: Time to last quantifiable concentration is based on last detectable concentration in the time curve.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h | 115.86 (33.4) | 113.79 (35.0) | 103.58 (41.0)

8. Primary Outcome: Time Between Dosing and Time of First Balovaptan Plasma Concentration (Tlag)
Description: Time between dosing and time of first balovaptan plasma concentration is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h | 0.2500 [0.0 to 1.5] | 0.2500 [0.0 to 0.5] | 0.2500 [0.0 to 0.5]

9. Primary Outcome: Apparent Clearance (Cl/F) of Balovaptan
Description: Apparent clearance is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
L/h | 11.51 (35.7) | 11.73 (36.3) | 11.26 (32.2)

10. Primary Outcome: Apparent Volume of Distribution (Vd/F) of Balovaptan
Description: Apparent volume of distribution is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
L | 422.7 (28.7) | 422.5 (33.4) | 429.4 (18.5)

11. Primary Outcome: Terminal Elimination Phase Half-Life (T1/2) of Balovaptan
Description: Terminal phase half-life expressed in time units is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 15
h | 25.44 (40.0) | 24.98 (47.0) | 27.26 (40.9)

12. Secondary Outcome: Maximum Plasma Concentration (Cmax) of M2 Metabolite
Description: Maximum plasma concentration of M2 Metabolite is estimated using non-compartmental methods. Observed peak analyte concentration obtained directly from the experimental data without interpolation, expressed in concentration units
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
ng/mL | 11.27 (27.0) | 11.44 (30.8) | 11.68 (30.1)

13. Secondary Outcome: Maximum Plasma Concentration (Cmax) of M3 Metabolite
Description: Maximum plasma concentration of M3 Metabolite is estimated using non-compartmental methods. Observed peak analyte concentration obtained directly from the experimental data without interpolation, expressed in concentration units
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
ng/mL | 15.96 (37.0) | 16.91 (40.8) | 16.85 (32.3)

14. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Esomeprazole
Description: Maximum plasma concentration of Esomeprazole is estimated using non-compartmental methods. Observed peak analyte concentration obtained directly from the experimental data without interpolation, expressed in concentration units
Time Frame: Samples at predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16
ng/mL | 1255.2 (36.9)

15. Secondary Outcome: Area Under the Concentration-Time Curve From Time Extrapolated to Infinity (AUC (0-inf)) of M2 Metabolite
Description: Area under the plasma concentration-time curve (time 0 to infinity) of M2 Metabolite is estimated using non-compartmental methods from the concentration-time profiles. Percent extrapolation less than or equal to 20% is required to obtain a reliable AUC0-inf.
Time Frame: as for outcome 1
Population: For one participant (Balovaptan 20 mg Fasted, Balovaptan 20 mg Fasted + Esomeprazole) AUC(0-inf)%extrap was > 20%, so AUC(0-inf) was not included in summary statistics. For one participant in Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fastedthere was no terminal phase, so AUC(0-inf) could not be calculated. One participant was discontinued in Period 3 with Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted after withdrawal of consent.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 15 | 14
h*ng/mL | 987.3 (27.5) | 998.5 (22.7) | 1087.7 (21.9)

16. Secondary Outcome: Area Under the Concentration-Time Curve From Time Extrapolated to Infinity (AUC (0-inf)) of M3 Metabolite
Description: Area under the plasma concentration-time curve (time 0 to infinity) of M3 Metabolite is estimated using non-compartmental methods from the concentration-time profiles. Percent extrapolation less than or equal to 20% is required to obtain a reliable AUC0-inf.
Time Frame: as for outcome 1
Population: Balovaptan 20 mg Fed: 3 participants were exluded from the analysis due to AUC(0-inf)%extrap > 20% Balovaptan 20 mg Fasted: 3 participants were exluded from the analysis due to AUC(0-inf)%extrap > 20% Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted: 4 participants were exluded from the analysis due to AUC(0-inf)%extrap > 20%. One additional participant was discontinued in Period 3 with Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted after withdrawal of consent.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 13 | 13 | 11
h*ng/mL | 1552.9 (26.2) | 1590.0 (26.9) | 1723.2 (26.5)

17. Secondary Outcome: Area Under the Concentration-Time Curve From Time Extrapolated to Infinity (AUC (0-inf)) of Esomeprazole
Description: Area under the plasma concentration-time curve (time 0 to infinity) of Esomeprazole is estimated using non-compartmental methods from the concentration-time profiles. Percent extrapolation less than or equal to 20% is required to obtain a reliable AUC0-inf.
Time Frame: Samples at predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose
Population: 3 participants were excluded from the analysis due to missing data. For one of those the value was excluded due to AUC(0-inf)%extrap > 20%.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 13
h*ng/mL | 4570.1 (48.7)

18. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to 24 Hours (AUC(0-24h)) of M2 Metabolite
Description: Area under the plasma concentration-time curve of M2 Metabolite from time 0 to 24 hours post-dose is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: Samples at predose, and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16 and 24 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h*ng/mL | 150.6 (38.3) | 180.1 (39.5) | 182.2 (35.9)

19. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to 24 Hours (AUC(0-24h)) of M3 Metabolite
Description: Area under the plasma concentration-time curve of M3 Metabolite from time 0 to 24 hours post-dose is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: Samples at predose, and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16 and 24 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h*ng/mL | 269.8 (40.9) | 325.1 (42.0) | 325.5 (34.1)

20. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of M2 Metabolite
Description: Area under the concentration-time curve (time 0 to time of last quantifiable concentration) of M2 Metabolite is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h*ng/mL | 897.6 (27.2) | 869.4 (26.9) | 873.9 (32.8)

21. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of M3 Metabolite
Description: Area under the concentration-time curve (time 0 to time of last quantifiable concentration) of M3 Metabolite is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h*ng/mL | 1389.6 (23.9) | 1462.8 (29.3) | 1384.3 (35.6)

22. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Esomeprazole
Description: Area under the concentration-time curve (time 0 to time of last quantifiable concentration) of Esomeprazole is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: Samples at predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16
h*ng/mL | 4014.9 (42.9)

23. Secondary Outcome: Time to Reach Cmax in Plasma (Tmax) of M2 Metabolite
Description: Time to maximum plasma concentration of M2 Metabolite is defined as first observed time to reach peak analyte concentration obtained directly from the experimental data without interpolation, expressed in time units and estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h | 36.00 [16.00 to 48.00] | 24.03 [16.00 to 48.00] | 36.00 [12.00 to 48.00]

24. Secondary Outcome: Time to Reach Cmax in Plasma (Tmax) of M3 Metabolite
Description: Time to maximum plasma concentration of M3 Metabolite is defined as first observed time to reach peak analyte concentration obtained directly from the experimental data without interpolation, expressed in time units and estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h | 20.01 [12.00 to 36.00] | 24.02 [4.00 to 36.00] | 16.00 [5.00 to 36.00]

25. Secondary Outcome: Time to Reach Cmax in Plasma (Tmax) of Esomeprazole
Description: Time to maximum plasma concentration of Esomeprazole is defined as first observed time to reach peak analyte concentration obtained directly from the experimental data without interpolation, expressed in time units and estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: Samples at predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose
Measure: Median (Full Range); unit: h
Arm/Group | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16
h | 2.00 [1.50 to 4.00]

26. Secondary Outcome: Last Quantifiable Concentration (Clast) of M2 Metabolite
Description: Last quantifiable concentration is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
ng/mL | 1.515 (30.0) | 1.739 (29.4) | 1.682 (82.8)

27. Secondary Outcome: Last Quantifiable Concentration (Clast) of M3 Metabolite
Description: Last quantifiable concentration is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
ng/mL | 2.211 (46.2) | 2.279 (55.4) | 2.837 (82.1)

28. Secondary Outcome: Last Quantifiable Concentration (Clast) of Esomeprazole
Description: Last quantifiable concentration is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: Samples at predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16
ng/mL | 133.3 (78.8)

29. Secondary Outcome: Time To the Last Quantifiable Concentration (Tlast) of M2 Metabolite
Description: Time to last quantifiable concentration is based on last detectable concentration in the time curve.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h | 155.3 (21.2) | 142.4 (25.2) | 142.4 (29.5)

30. Secondary Outcome: Time To the Last Quantifiable Concentration (Tlast) of M3 Metabolite
Description: Time to last quantifiable concentration is based on last detectable concentration in the time curve.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
h | 192.0 (0.0) | 192.0 (0.0) | 168.7 (23.1)

31. Secondary Outcome: Time To the Last Quantifiable Concentration (Tlast) of Esomeprazole
Description: Time to last quantifiable concentration is based on last detectable concentration in the time curve.
Time Frame: Samples at predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16
h | 8.002 (0.1)

32. Secondary Outcome: Terminal Elimination Phase Half-Life (T1/2) of M2 Metabolite
Description: as for outcome 11
Time Frame: as for outcome 1
Population: For one participant in Balovaptan 20 mg Fasted and one participant in Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted AUC(0-inf)%extrap was > 20%, so T1/2 were not included in summary statistics. For one additional participant in Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted there was no terminal phase, so AUC(0-inf) and T1/2 could not be calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 15 | 14
h | 38.99 (29.2) | 37.81 (30.7) | 39.19 (22.7)

33. Secondary Outcome: Terminal Elimination Phase Half-Life (T1/2) of M3 Metabolite
Description: as for outcome 11
Time Frame: as for outcome 1
Population: For 3 subjects in Balovaptan 20 mg Fed, 3 subjects in Balovaptan 20 mg Fasted and 4 subjects in Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted AUC(0-inf)%extrap was > 20%, so AUC(0-inf) were not included in summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 13 | 13 | 11
h | 57.40 (17.3) | 59.30 (17.6) | 57.81 (19.2)

34. Secondary Outcome: Terminal Elimination Phase Half-Life (T1/2) of Esomeprazole
Description: as for outcome 11
Time Frame: Samples at predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose
Population: For one participant AUC(0-inf)%extrap was > 20%, so T1/2 was not included in summary statistics. For 2 participants, there was no terminal phase, so T1/2 could not be calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 13
h | 1.590 (29.2)

35. Secondary Outcome: Percentage of Patricipants With Adverse Events (AEs)
Time Frame: Randomization to end of study (up to approximately 7 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
Participants | 1 | 1 | 1

36. Primary Outcome: Terminal Phase Rate Constant (λz) of Balovaptan
Description: Terminal phase rate constant is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
/h | 0.0272 (33.3) | 0.0278 (37.5) | 0.0263 (30.3)

37. Secondary Outcome: Terminal Phase Rate Constant (λz) of M2 Metabolite
Description: Terminal phase rate constant is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Population: For one participant there was no terminal phase, so they are excluded form the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 15
/h | 0.0178 (30.3) | 0.0174 (31.9) | 0.0171 (25.5)

38. Secondary Outcome: Terminal Phase Rate Constant (λz) of M3 Metabolite
Description: Terminal phase rate constant is estimated using non-compartmental methods from the concentration-time profiles.
Time Frame: as for outcome 1
Population: For one participant there was no terminal phase, so they are excluded form the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /h
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 15
/h | 0.0112 (22.1) | 0.0107 (24.8) | 0.0107 (25.2)

39. Secondary Outcome: Terminal Phase Rate Constant (λz) of Esomeprazole
Description: as for outcome 11
Time Frame: Samples at predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose
Population: For two participants there was no terminal phase, so they are excluded form the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /h
Arm/Group | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 14
/h | 0.4197 (30.1)

40. Primary Outcome: Plasma Concentrations of Balovaptan
Description: Amount of Balovaptan in a given volume of plasma.
Time Frame: as for outcome 1
Population: Number of analyzed participants reflects number of participants whose samples were available at given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
ng/mL
  Predose | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL)
  0.25 Hrs Postdose | 3.90 (246.8) | 2.46 (136.0) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL)
  0.5 Hrs Postdose | 8.89 (235.7) | 21.26 (117.5) | 8.40 (129.8)
  1 Hrs Postdose | 17.76 (113.0) | 63.58 (60.9) | 44.78 (70.8)
  1.5 Hrs Postdose | 20.08 (88.2) | 66.54 (47.4) | 49.82 (52.7)
  2 Hrs Postdose | 27.47 (77.0) | 70.75 (32.9) | 62.24 (37.0)
  2.5 Hrs Postdose | 32.90 (73.0) | 66.40 (33.4) | 63.44 (32.1)
  3 Hrs Postdose | 41.92 (73.6) | 63.60 (29.7) | 66.26 (29.8)
  3.5 Hrs Postdose | 45.68 (60.4) | 60.63 (31.2) | 64.70 (34.5)
  4 Hrs Postdose | 51.84 (50.2) | 59.58 (27.9) | 63.95 (31.5)
  5 Hrs Postdose | 60.59 (36.5) | 59.56 (27.4) | 61.45 (35.4)
  6 Hrs Postdose | 56.91 (34.6) | 49.69 (28.3) | 54.51 (31.1)
  8 Hrs Postdose | 51.07 (30.7) | 44.58 (30.0) | 48.05 (30.5)
  12 Hrs Postdose | 39.18 (27.4) | 34.74 (32.9) | 35.91 (31.8)
  16 Hrs Postdose | 33.17 (38.5) | 28.88 (37.5) | 30.85 (37.1)
  24 Hrs Postdose | 25.43 (42.7) | 22.95 (43.6) | 25.95 (37.2)
  36 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  36 Hrs Postdose | 14.94 (57.1) | 13.92 (55.4) | 15.13 (50.1)
  48 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  48 Hrs Postdose | 9.75 (70.5) | 10.70 (7.376) | 12.15 (6.794)
  72 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  72 Hrs Postdose | 4.47 (90.2) | 4.28 (97.8) | 5.04 (64.0)
  96 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  96 Hrs Postdose | 2.68 (112.0) | 2.86 (125.0) | 2.98 (91.4)
  144 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  144 Hrs Postdose | 2.38 (186.5) | 2.45 (204.4) | 2.57 (198.5)
  192 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  192 Hrs Postdose | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL)

41. Secondary Outcome: Plasma Concentrations of M2 Analyte
Description: Amount of M2 Analyte in a given volume of plasma.
Time Frame: as for outcome 1
Population: Number of analyzed participants reflects number of participants whose samples were available at given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
ng/mL
  Predose | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL)
  0.25 Hrs Postdose | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL)
  0.5 Hrs Postdose | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL)
  1 Hrs Postdose | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | 3.081 (62.2) | 2.649 (95.5)
  1.5 Hrs Postdose | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | 3.421 (57.2) | 2.690 (72.6)
  2 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  2 Hrs Postdose | 2.021 (97.7) | 3.637 (45.6) | 3.019 (54.9)
  2.5 Hrs Postdose | 2.236 (83.3) | 3.724 (48.8) | 3.502 (46.4)
  3 Hrs Postdose | 2.714 (80.0) | 4.293 (49.9) | 3.878 (43.2)
  3.5 Hrs Postdose | 2.780 (75.7) | 4.724 (49.2) | 4.217 (44.5)
  4 Hrs Postdose | 3.208 (65.5) | 4.860 (49.1) | 4.749 (41.1)
  5 Hrs Postdose | 3.756 (60.5) | 5.696 (47.9) | 5.471 (44.8)
  6 Hrs Postdose | 4.158 (50.9) | 5.797 (50.0) | 5.775 (39.8)
  8 Hrs Postdose | 5.223 (48.9) | 6.550 (46.6) | 6.512 (40.8)
  12 Hrs Postdose | 6.921 (40.4) | 7.889 (39.5) | 8.426 (42.9)
  16 Hrs Postdose | 8.384 (39.7) | 9.207 (40.9) | 9.563 (34.2)
  24 Hrs Postdose | 10.123 (29.4) | 10.928 (30.9) | 10.887 (33.0)
  36 Hrs Postdose | 10.509 (29.6) | 10.519 (27.4) | 11.409 (26.9)
  48 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  48 Hrs Postdose | 9.383 (28.2) | 9.134 (25.8) | 10.191 (26.8)
  72 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  72 Hrs Postdose | 6.576 (30.7) | 5.998 (27.5) | 27.5 (23.5)
  96 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  96 Hrs Postdose | 4.050 (41.6) | 3.748 (32.9) | 4.450 (27.5)
  144 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  144 Hrs Postdose | 2.033 (64.7) | 2.139 (71.9) | 2.107 (45.2)
  192 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  192 Hrs Postdose | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL)

42. Secondary Outcome: Plasma Concentrations of M3 Analyte
Description: Amount of M3 Analyte in a given volume of plasma.
Time Frame: as for outcome 1
Population: Number of analyzed participants reflects number of participants whose samples were available at given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
ng/mL
  Predose | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL)
  0.25 Hrs Postdose | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL)
  0.5 Hrs Postdose | NA (NA) — Below Quantifiable Limit (< 1.00 ng/mL) | 5.006 (118.0) | 3.172 (127.1)
  1 Hrs Postdose | 2.347 (138.4) | 7.812 (60.6) | 5.556 (78.9)
  1.5 Hrs Postdose | 3.787 (95.1) | 8.928 (59.6) | 6.705 (62.6)
  2 Hrs Postdose | 5.211 (83.0) | 10.157 (46.8) | 8.859 (55.8)
  2.5 Hrs Postdose | 5.520 (83.5) | 10.539 (47.9) | 9.853 (45.8)
  3 Hrs Postdose | 6.616 (85.9) | 10.980 (48.6) | 10.887 (39.4)
  3.5 Hrs Postdose | 5.985 (78.0) | 11.369 (50.8) | 11.316 (41.2)
  4 Hrs Postdose | 6.408 (71.4) | 12.160 (50.8) | 11.969 (38.0)
  5 Hrs Postdose | 8.901 (58.8) | 13.241 (41.5) | 12.998 (46.7)
  6 Hrs Postdose | 9.691 (59.8) | 12.831 (47.9) | 13.442 (39.6)
  8 Hrs Postdose | 11.157 (47.8) | 13.875 (48.4) | 13.762 (40.4)
  12 Hrs Postdose | 12.697 (5.7063) | 14.296 (39.7) | 14.287 (36.3)
  16 Hrs Postdose | 14.113 (40.9) | 15.145 (41.6) | 15.049 (30.1)
  24 Hrs Postdose | 14.388 (33.4) | 15.061 (39.7) | 16.092 (29.9)
  36 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  36 Hrs Postdose | 13.626 (26.4) | 14.148 (29.7) | 13.793 (27.7)
  48 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  48 Hrs Postdose | 11.665 (26.4) | 11.470 (29.0) | 12.966 (27.3)
  72 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  72 Hrs Postdose | 8.108 (28.3) | 8.129 (31.3) | 9.023 (25.2)
  96 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  96 Hrs Postdose | 6.066 (31.6) | 6.111 (42.4) | 6.653 (34.1)
  144 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  144 Hrs Postdose | 3.525 (45.5) | 3.747 (45.7) | 3.957 (45.2)
  192 Hrs Postdose: number analyzed (Participants) | 16 | 16 | 15
  192 Hrs Postdose | 2.211 (46.2) | 2.279 (55.4) | 2.569 (54.2)

43. Secondary Outcome: Plasma Concentrations of Esomeprazole
Description: Amount of Esomeprazole in a given volume of plasma.
Time Frame: Samples at predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose
Population: Number of analyzed participants reflects number of participants whose samples were available at given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
Number analyzed (Participants) | 16
ng/mL
  Predose | NA (NA) — Below Quantifiable Limit (< 2.00 ng/mL)
  0.25 Hrs Postdose | NA (NA) — Below Quantifiable Limit (< 2.00 ng/mL)
  0.5 Hrs Postdose | NA (NA) — Below Quantifiable Limit (< 2.00 ng/mL)
  1 Hrs Postdose | 171.8 (171.5)
  1.5 Hrs Postdose | 242.6 (102.8)
  2 Hrs Postdose | 697.1 (66.2)
  3 Hrs Postdose | 984.4 (36.1)
  4 Hrs Postdose | 770.7 (34.7)
  6 Hrs Postdose | 336.6 (59.8)
  8 Hrs Postdose | 133.3 (78.8)

ADVERSE EVENTS:
Time Frame: From baseline to end of study (up to approximately 7 weeks)
Arm/Group | Balovaptan 20 mg Fed | Balovaptan 20 mg Fasted | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 1/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balovaptan 20 mg Fed (N=16) | Balovaptan 20 mg Fasted (N=16) | Balovaptan 20 mg Fasted + Esomeprazole 40 mg Fasted (N=16)
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT04156646/Prot_SAP_000.pdf